CLINICAL TRIAL: NCT00783627
Title: Evaluation of Angiogenic Potential in Sickle Cell Disease. CARACTERIZATION of Endothelial Progenitor Cells
Brief Title: Sickle Cell Disease and Endothelial Progenitor Cells (EPCs)
Acronym: DREPANOPEC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Aucan, Department Clinical Research of Developpement
Other Study IDs: P 050310
Record Dates: First submitted 2008-10-15; First posted 2008-11-03 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Sickle Cell Anemia
Keywords: Endothelium; progenitors; stem cells; sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Cerebral Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patient with sickle cell disease
  Interventions: Procedure: Angiography
- 2: Healthy volunteers

INTERVENTIONS:
Procedure: Angiography — Angiography done at the J1 visit
  Groups: 1

SUMMARY:
Sickle Cell Disease (SCD) is the most prevalent genetic disease of haemoglobin.The underlying abnormality in the red blood cell (RBC) of SCD is the presence of abnormal sickle cell hemoglobin (HbS), which, when deoxygenated, becomes relatively insoluble, forms aggregates with other hemoglobin molecules within the RBC and causes rigid deformation of the cell. Acute pain vaso-occlusive crisis, strokes and acute chest syndrome are the main acute complications, sometimes life-threatening, often leading to organic and functional squeal. Although the common SS form of SCD is a unique gene disorder, the range of the clinical severity is remarkably wide and striking, suggesting that clinical polymorphism is due to modifier genes and environmental factors.Most of the research efforts have been focused on the biology of haemoglobin and of the red cells. Meanwhile, the complex pathophysiology of SCD is undoubtedly influenced by the many physiologic functions of the vascular wall. In line with this hypothesis are several reports of increased circulating levels of endothelium-derived surface molecules in SCD patients suggesting marked endothelial stress in SCD. Similarly, other processes that involve the endothelium, such as leukocyte adhesion and activation, may play a role in vascular occlusion. This accumulation of data raises the unanswered question of the mechanisms of endothelium maintenance and regeneration in SCD. Through these mechanisms, it is likely that function or dysfunction of the vascular endothelium contributes to the overall vascular pathobiology of this disease, which includes recurrent vaso-occlusions, stroke, leg ulcers, chronic organ ischemic damages, and neovascularizing retinopathy that affect nearly one-half (48%) of the surviving patients by the fifth decade.Thus, our groups have combined their respective clinical and biological expertises to test the hypothesis that SCD is a condition of specific endothelial stress and dysfunction upon chronic and Paracystic abnormal interactions with circulating cells and abnormal oxygen delivery to tissues. Specifically, we hypothesize that chronic endothelial stress with detachment of activated endothelial cells require increases mobilisation of the Endothelial Progenitor Cells (EPCs) that maintain endothelial homeostasis to avoid major thromboembolic events and vasospasm. Inappropriate mobilisation or maturation of the EPCs in SCD may participate to the severity of the disease.

DETAILED DESCRIPTION:
In the bone marrow, a reservoir of EPCs does exist, which can be mobilized into circulation when needed, for example during ischemia, a situation which may occur in sickle cells disease. These cells are able to reach distant targets and to participate to the neovascularisation processes necessary for tissue and vascular healing. Conversely, abnormalities of the maturation, mobilization or homing processes would contribute to the thrombotic and ischemic risks associated to ischemia. Furthermore, vascular stress such that encountered in SCD leads to the detachment of endothelial cells from the vessels. The number of detached mature circulating endothelial cells (CEC) seems to be related to vascular hurting. The balance between EPCs and CECs would thus be informative of the vascular condition in patients during the progression of the disease. A relatively high level of EPCs would indicate a prominence of a healing neoangiogenesis or vasculogenesis process, while increasing levels of CECs would be indicative severe progression of the disease. Our studies and those published by others indicate that the number of EPCs in peripheral blood is tightly regulated. Indeed, mediators of inflammation could participate to EPC mobilization and to their recruitment to the diseased areas by local activation of the vascular endothelium. In this context, sickle cells disease provokes transient occlusion episodes, leading to a situation of chronic ischemia in different organs, sometimes with acute episodes. This suggests defect of the maintenance of the vascular integrity in these target organs.Within this project, we will compare the number of EPCs and CECs in 25 SCD patients and 25 normal individuals in search of a correlation with the severity of the disease. SCD patients with potential confounding factors that may alter endothelial physiology (drugs, blood transfusions, hydroxyurea therapy) are excluded. In addition, we will analyse and compare in culture and in vivo the phenotypic and functional characteristics of EPCs obtained from patients and controls. We have a working bilateral hypothesis, since we do not know whether SCD subjects have appropriate angiogenic balance (high EPCs/CEC ratio with functional EPCs) to face the situation of endothelial activation and tissue hypoxia induced by SCD. Therefore, we will quantitatively and qualitatively study several distinct biological steps:1. Evaluate the number of colonies generated by the EPCs in culture and their kinetics of appearance in patients (major end point)2. Enumerate EPCs and CECs by flow cytometry using a specific set of markers (CD133, CD146, KDR).3. Measure of the plasma concentrations of PlGF, VEGF, EPO, ET-1, modulators of angiogenesis.4. Test of correlations between these respective characteristics of EPCs with clinical vascular abnormalities of the disease (retinopathy assessed by angiography, nephropathy, leg ulcers) and severity of vaso-occlusive crisis assessed by number and length of hospitalizations during the previous year and during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 yo
* SS genotype if patient
* Absence of relative with sickle cell anemia if healthy volunteer.
* Affiliated to the national health insurance benefit
* Signature of Informed consent form
* oral contraceptive regiment with micro or mini estro-progestative (women)

Exclusion Criteria:

* present or past (or interrupted for less than 3 months) therapy with hydroxyurea
* Present or recent blood transfusion and/or exchange (in the past 3 months)
* SC genotype (patients)- BMI > 30 kg/m2
* Positive serodiagnosis for HIV, HVB, HVC
* Know allergy to fluorescein (patients)
* Hemoglobin < 7.5 g/dL
* Pregnancy confirmed by Beta-HCG test in plasma
* Menopause
* Extreme difficulty for adequate venous puncture
* Smoking for the last month.
* ALAT or ASAT > 2 x N
* Hypercholesterolemia (cholesterol total > 2.,2g/L or 6.55 mmol/L),
* Treatment by statin
* Diabetes (fasting blood glucose level equal or superior to 6,1 mmol/L)
* Hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sickle cell patient : followed by the participating center. Healthy volunteers : matched on sex, age and BMI with the patients.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Measure the relative levels of endothelial progenitors (EPCs) derived from cultured mononuclear cells in patients and carefully matched healthy subjects at day 0 and after 6 months later (number of endothelial cells colony forming units). | at day 0 and 6 months

SECONDARY OUTCOMES:
Comparison of the number of circulating EPCs and CECs by FACS. The blood mononuclear cell fraction are depleted from all the haematopoietic cells using a depletion magnetic bead column. The lineage minus population is then subjected to a triple labelling | at day 1 and at 6 months
Correlations tests will be performed between these markers and markers of clinical severity (retinopathy, leg ulcers, number of vaso-occlusive events in the past year, microalbuminuria, leukocyte count, HbF level). | at day 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Louis THARAUX, MDPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Tenon, Assistance Publique Hôpitaux de Paris, Paris, France